CLINICAL TRIAL: NCT06571773
Title: Evaluation of Astigmatism-correcting IOL Combined With Tension Ring on Postoperative Visual Quality and Rotational Stability of IOLs in Patients With Cataract Combined With High Myopia
Brief Title: Evaluation of Toric Intraocular Lens(IOL) Combined With Capsular Tension Ring(CTR) in Patients With Cataract Combined With High Myopia
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Sun Yilin, Resident Physician, Shanghai 10th People's Hospital
Other Study IDs: SHISY-LYZX-217
Record Dates: First submitted 2024-08-23; First posted 2024-08-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2024-08

CONDITIONS: Cataract; Astigmatism; Intraocular Lens Rotation
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CTR group: This group include the patients with the usage of CTR
  Interventions: Procedure: intraoperative implantation of Capsular Tension Ring
- control group: This group include the patients without the usage of CTR
  Interventions: Procedure: none intraoperative implantation of CTR

INTERVENTIONS:
Procedure: intraoperative implantation of Capsular Tension Ring — The Capsular Tension Ring(ACPi-11; Bausch + Lomb, Rochester, New York, USA) is a device made of PMMA with blunt-tipped eyelets at its ends. It can be inserted at any point during cataract surgery, following the creation of a strong anterior capsulotomy via capsulorhexis
  Groups: CTR group
Procedure: none intraoperative implantation of CTR — the surgeon did a surgery without the intraoperative implantation of CTR
  Groups: control group

SUMMARY:
The objective of this study is to evaluate the postoperative visual quality and IOL stability in patients with cataracts and high myopia who have undergone surgery using astigmatism-correcting IOLs in conjunction with tension rings.It is a non-randomised retroprospective cohort study. Patients with high axial myopia (AL ≥ 26 mm) who underwent cataract phacoemulsification combined with toric IOL(Acrysof SN6ATY IQ toric IOL, Alcon, Alcon Laboratories, Fort Worth, Texas, USA) implantation from October 2020 to September 2023 at the Shanghai Tenth People's Hospital are selected. According to the usage of CTR, all patients will be divided into CTR group and control group, with a minimum follow-up of 3 months.Each patient underwent a comprehensive preoperative examination and ophthalmological examinations at the outpatient clinic 1 day, 1 week, 1 month, and 3 months postoperatively.Statistical analysis will be conducted using SPSS 26.0 statistical software.

DETAILED DESCRIPTION:
Preoperative examination:Each patient underwent a comprehensive preoperative examination, which included evaluation of uncorrected visual acuity (UCVA), best corrected visual acuity (BCVA), corneal endothelial cells (CECs), axial length, corneal curvature, and corneal topography using subjective optometry, slit-lamp microscopy, funduscopic examination, intraocular pressure measurements, B-scan ultrasound of the eye, and corneal topography(Pentacam HR, OCULUS Optikgerate, Wetzlar, Germany), as well as other relevant parameters. Visual acuity was measured using a standard logarithmic visual acuity chart. Biometry of the operative eye was performed by a specialized technician using an IOL Master (IOLMaster 700, Carl Zeiss Meditec, Jena, Germany), and the Barret's formulaⅡ was applied to calculate the equivalent spherical equivalent (SE) of the toric IOL. The information was inputted into an online calculator (www.acrysoftoriccalculator.com) provided by Alcon to determine the necessary IOL refraction and axial position.

Surgery:The patients received tobramycin dexamethasone eye drops four times one day before surgery. Prior to surgery, the IOL axial position, the diameter size of continuous curvilinear capsulorhexis (CCC), and the incision position were measured and marked using the Image Guided System(VERION Reference Unit, Alcon GPS-WaveLight GmbH, Rheinstrasse, Germany). The pupil was dilated with compound tropicamide drops to a diameter of at least 8mm. The surgery was performed by an experienced surgeon following a standardized procedure. The surgical procedure was as follows: Proparacaine hydrochloride eye drops (ALCAINE, S.A.Alcon-Couvreur N.V., Belgium) were used to provide surface anaesthesia. The conjunctival sac was rinsed with 1% povidone-iodine. Afterwards, a 2.2-mm corneal incision and a 15° stab knife auxiliary incision were made under the guidance of digital navigation system. Inserting the viscoelastic into the anterior chamber and applying a continuous circular capsulorhexis method, a complete hydro dissection was performed. The lens nucleus was removed using ultrasonic emulsification, follow by aspirating the excess cortex and polishing the capsule. After propping up the capsular bag with viscoelastic, the intraocular lens (IOL) was implanted through the main incision (the CTR would be implanted before the IOL implantation). After suctioning off the viscoelastic, the IOL was adjusted to the predetermined axis under navigation guidance. Finally, the incision was hydrated. Tobramycin dexamethasone eye drops were used for 2 weeks postoperatively in all cases.

Postoperative management:All patients underwent ophthalmological examinations at the outpatient clinic 1 day, 1 week, 1 month, and 3 months postoperatively. The examinations included uncorrected distance visual acuity, intraocular pressure examination, subjective optometry, slit lamp microscopy, and SS-OCT (CASIA2, Tomey Corporation, Nagoya, Japan). The surgeon, using the same slit lamp microscope and a narrow band of light, measured the IOL axial position after the patients' pupils were fully dilated with compound tropicamide eye drops. The rotation degree was calculated as the absolute difference between the axial positions of the check and target.

ELIGIBILITY:
Inclusion Criteria:

* Cataract ultrasonic emulsification aspiration with one-stage implantation of astigmatic IOL at the Shanghai Tenth People's Hospital from October 2020 to September 2023;
* Ocular axial length ≥26.00mm;
* Completion of outpatient follow up for more than 3 months.

Exclusion Criteria:

* irregular corneal astigmatism, iris abnormalities, and pupil distortion;
* history of previous corneal or intraocular surgery;
* previous ocular diseases such as uveitis, retinopathy, macular degeneration, glaucoma, and keratoconus;
* postoperative posterior capsule rupture, and suspensory ligament dissociation of greater than 1 quadrant;
* corneal endothelial cell counts of less than 2000 cells/mm2.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cataract ultrasonic emulsification aspiration with one-stage implantation of astigmatic IOL at the Shanghai Tenth People's Hospital from October 2020 to September 2023
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative IOL rotation degree | 3 months
  The surgeon, using the same slit lamp microscope and a narrow band of light, measured the IOL axial position after the patients' pupils were fully dilated with compound tropicamide eye drops

CONTACTS AND LOCATIONS:
Overall Officials: Yili Sun, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China